CLINICAL TRIAL: NCT05395533
Title: A Multicenter, Single-arm, Dose-escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Effectiveness of TRS005 in Patients With Relapsed or Refractory CD20-positive B-NHL
Brief Title: A Phase 1 Study of TRS005 in Patients With R/R CD20-positive B-NHL.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Teruisi Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRS00501001
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: CD20-positive B-cell Non-Hodgkin Lymphoma
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Recombinant CD20 monoclonal antibody-MMAE conjugte for injection (TRS005) (Experimental): To evaluate the safety and tolerability of TRS005 in patients with recurrent or refractory CD20-positive B-cell non-Hodgkin's lymphoma with treatment at one or more times, and to recommend the dose for phase II clinical trials (RP2D).
  Interventions: Drug: Recombinant CD20 monoclonal antibody-MMAE conjugte for injection

INTERVENTIONS:
Drug: Recombinant CD20 monoclonal antibody-MMAE conjugte for injection — The dose of the enrolled subjects was increased according to the following 6 dose groups: 0.1mg/kg, 0.5mg/kg, 1.0mg/kg, 1.5mg/kg, 1.8mg/kg, and 2.1mg/kg.
  Other Names: TRS005

SUMMARY:
This trial is a multicenter, open, single arm, dose increasing and extended clinical trial. The dose was increased according to the "3 + 3" rule. Patients with recurrent or refractory CD20 positive B-cell non-Hodgkin's lymphoma were selected to evaluate the safety, tolerance (DLT, MTD) and pharmacokinetic (PK) characteristics of TRS005 by intravenous drip.

DETAILED DESCRIPTION:
The subjects were screened and examined according to the protocol before enrollment. The dose of the enrolled subjects was increased according to the following 6 dose groups: 0.1mg/kg, 0.5mg/kg, 1.0mg/kg, 1.5mg/kg, 1.8mg/kg, 2.1mg/kg. The incremental process is divided into groups according to the principle of 3 + 3 dose increment. The subjects randomly receive intravenous drip of TRS005 in chronological order. Each subject first carries out a single dose study, and then carries out multiple continuous doses. The first dose is given once in D1. After 21 days of observation, it is decided whether to continue multiple continuous doses according to the situation. They are given once in C2D1, C3D1, C4D1, C5D1, C6D1, or more cycles respectively, and received treatment until progressive disease or unacceptable toxicity. During the dose escalation process, the investigators will perform dose expansion according to the clinical benefits of different dose groups.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CD20-positive B-cell non-Hodgkin lymphoma;
2. Relapse or refractory after receiving at least 2 standard treatment regimens;（Definition of refractory: Patients who did not reach PR in two cycles or CR in four cycles）;
3. At least 1 measurable tumor lesion, the maximum transverse diameter of the intranodal lesion should be > 1.5 cm and that of the extranodal lesion should be > 1.0 cm; CLL/SLL patients have treatment indications according to iwCLL 2018 guidelines;
4. Previously received anti-tumor treatment (such as radiotherapy, chemotherapy, hormone therapy, biotherapy, immunotherapy) at least 28 days before the first administration of this study; chemotherapy and hormono therapy should be at least 14 days before the first administration of this study; Chinese medicine anti-tumor treatment should be at least 7 days before the first administration of this study
5. The toxicity of previous anti-tumor treatment has been restored to ≤ grade 1 as defined by NCI-CTCAE v5.0 (except for alopecia; see Inclusion Criterion 6 for hemoglobin and renal function)；
6. The laboratory test results must meet the following requirements: (It is not allowed to give any blood components, short acting cell growth factor, albumin, etc., within 7 days before laboratory examination; long acting cell growth factor is not allowed to be given within the first 14 days):

   * Hematology: Absolute neutrophil count (ANC) ≥ 1.5×109/L, platelets (PLT) ≥ 90×109/L, hemoglobin (HGB) ≥ 90 g/L;
   * Liver function: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal, total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal, (AST and/or ALT ≤ 5 times the upper limit of normal are allowed in patients with liver involvement);
   * Renal function: Serum creatinine (Cr) ≤ 2 times the upper limit of normal;
   * Coagulation function: (patients who have not received anticoagulant treatment before enrollment) International normalized ratio (INR) ≤ 1.5 times the upper limit of normal and activated partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of normal;
   * Pulmonary function test for patients with previous lung underlying disorders: measured/predicted value of vital capacity (VC) ≥ 60%, or diffusing capacity of the lungs for carbon monoxide (DLCO) ≥ 50% of predicted value;
7. ≥ 18 years , gender is not limited;
8. ECOG performance status 0-1;
9. Life expectancy of greater than 3 months;
10. Female and male patients of childbearing age and their spouses are willing to carry out adequate contraception throughout the study period, and female patients of childbearing age must have negative serum pregnancy test within 7 days before the first administration;
11. Patients voluntarily agree to participate in the study and to sign the informed consent form.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded:

1. A clear history of drug allergy, and a history of ingredient allergy to heterogeneous proteins, biological agents or test drugs;
2. Active hepatitis B or C, or human immunodeficiency virus (HIV) antibody positive;
3. Those who are positive for syphilis antibodies and confirmed to be unresolved;
4. Tumor-infiltrating diseases of the central nervous system;
5. Accompanied by peripheral or central nervous system diseases;
6. Investigator-assessed diabetes uncontrolled by drug therapy;
7. Uncontrollable or symptomatic pleural/abdominal/pelvic effusion or pericardial effusion;
8. Patients with other malignancies within the past 5 years;
9. With active autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, etc.);
10. Accompanied by the following serious cardiovascular diseases or central nervous system diseases:

    1. Myocardial infarction in nearly 6 months of screening period;
    2. Unstable angina pectoris in the screening period of nearly 3 months;
    3. Cardiac insufficiency (cardiac function grade ≥ NYHA class II);
    4. Severe arrhythmia (e.g., persistent ventricular tachycardia, ventricular fibrillation);
    5. Prolonged QTc interval (male > 450 ms, female > 470 ms);
    6. Second or third degree heart block;
    7. Drug-poorly controlled hypertension (systolic blood pressure > 160mmHg or diastolic blood pressure > 100mmHg);
    8. Cerebrovascular accident (CVA) or transient ischemic attack (TIA), etc., within 6 months before the administration.
11. Other serious diseases, including but not limited to active peptic ulcer, active hemorrhage, venous thromboembolic event (VTE) and severe interstitial lung disease;
12. Accompanied by other serious diseases and serious active infections (such as pneumonia, active tuberculosis, etc.);
13. Received hematopoietic growth factor treatment within 1 week prior to first administration, including colony stimulating factor, interleukin or blood transfusion;
14. The dosage of steroid hormone (prednisone phase equivalent) used greater than 20mg/ day within 1 month prior to first administration for more than 14 consecutive days or immunosuppressive treatment;
15. Various vaccines were inoculated within 1 month prior to first administration;
16. Major surgery (except diagnostic biopsy) within 1 month prior to first administration;
17. Patients who received autologous stem cell transplantation within 2 months prior to first administration;
18. Patients who have received allogeneic stem cell transplantation in the past;
19. Patients with infusion reaction above grade III after previous monoclonal antibody treatment;
20. Participate in clinical trials of other drugs or medical devices within 1 month prior to first administration;
21. Patients previously treated with CAR-T;
22. Investigators assessed as unsuitable to participate in this study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Toxicity | Cycle 1(Days 1-21)
  DLTs were defined as specific events which occurred in the 21-day DLT evaluation period of the dose escalation part, except any events that were clearly due to underlying disease or extraneous causes. The grading and severity of events were based on the guidelines provided in the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
MTD，Maximum Tolerated Dose | Cycle 1(Days 1-21)
  After the dose increment is completed, the incidence of DLT in each dose group is summarized and analyzed. The highest dose group closest to 1 / 3 of the preset incidence of DLT is MTD
Number of Participants With Treatment-emergent Adverse Event (TEAE) | Baseline up to approximately 5 years
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. AEs were reported based on the national cancer institute common terminology criteria for AEs, Version 5.0 (NCI-CTCAE, v5.0). Reported are the number of subjects with AEs, Grade 3-5 AEs, and Serious Adverse Events (SAEs).

SECONDARY OUTCOMES:
Number of Participants With ADA/Nab | Baseline up to approximately 5 years
  Evaluate the changes of anti drug antibody and neutralizing antibody produced by the subjects.
ORR, overall response rate | Baseline up to approximately 5 years
  Summarize the number and percentage of objective remission (Complete remission (CR) or Partial remission (PR))
DOR, duration of response | Baseline up to approximately 5 years
  DOR was defined as the time from the documentation of first tumor response (CR or PR) to disease progression or death.
PFS, progression-free survival | Baseline up to approximately 5 years
  PFS was defined as the time between start of treatment and the first documentation of progression, or death.
OS, overall survival | Baseline up to approximately 5 years
  OS was defined as the time between the start of treatment and death from any cause.
Cmax | At the day3/day5/day8/day15 in cycle 1and 4；and at the first day of Cycle 1-5 (each cycle is 21 days)
  Peak concentration. Obtained directly from the measured data of blood drug concentration-time.
AUC0-t | At the day3/day5/day8/day15 in cycle 1and 4；and at the first day of Cycle 1-5 (each cycle is 21 days)
  Area under the curve from zero to the lowest detectable plasma concentration. Calculated by linear trapezoidal rule:
  AUC(i, i+1)=(Ti+1-Ti)(Ci+Ci+1)/2, AUC 0-t is the sum of all AUC (I, I + 1).
AUC0-∞ | At the day3/day5/day8/day15 in cycle 1and 4；and at the first day of Cycle 1-5 (each cycle is 21 days)
  Area under the curve extrapolated from zero to infinity time. AUC0-∞=AUC0-t+Ct/λ z(Ct is the last measurable plasma concentration)
Tmax | At the day3/day5/day8/day15 in cycle 1and 4；and at the first day of Cycle 1-5 (each cycle is 21 days)
  Peak time. Obtained directly from the measured data of blood drug concentration-time.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (6):
- China (6):
  - Chinese Academy of Medical Sciences, Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center (SYSUCC), Guangzhou, Guangdong
  - Henan Cancer Hospital (Affiliated Cancer Hospital of Zhengzhou University), Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Tianjin Medical University Cancer Institute & Hospital (TMUCIH), Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No